CLINICAL TRIAL: NCT04995731
Title: Risk Assessment of Endometrial Hyperplasia and Endometrial Cancer: Development and Validation of Clinical-ultrasound Based Scoring System(A Cross Sectional -Validation Study)
Brief Title: Risk Assessment of Endometrial Hyperplasia and Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan Tarek Sayed, assistant lecturer of obstetrics and gynecology, Faculty of medicine, Assiut University
Other Study IDs: AssiutNT
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Endometrial Cancer
Keywords: endometrial hyperplasia
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Endometrial sampling either through hysteroscopy or dilatation and curettage operation (D, C) or histopathological evaluation of biopsy specimens obtained by hysterectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with pre or peri-menopausal abnormal uterine bleeding or post menopausal bleeding: Eligible women presenting to Women's Health hospital with pre or peri-menopausal AUB or PMB will be prospectively enrolled after obtaining their informed consent. AUB will be deﬁned by symptoms of heavy menstrual bleeding, inter-menstrual bleeding, meno-metrorrhagia, irregular menses, or other AUB among women aged ≥40 years who are not in menopause. Peri-menopausal bleeding will be defined as vaginal bleeding after 6 months of menopause after the age of 40 years. Postmenopausal status will be defined as the absence of menstruation for at least 12 months after the age of 40 years, where any pathological condition of amenorrhea is excluded.
  Interventions: Behavioral: Information about clinical risk factors for endometrial cancer and endometrial hyperplasia (EH); Procedure: transvaginal ultrasound examination

INTERVENTIONS:
Behavioral: Information about clinical risk factors for endometrial cancer and endometrial hyperplasia (EH) — Bleeding type, age, race, parity, early menarche or late menopause, body mass index, body composition, hypertension, type II diabetes, anovulation, polycystic ovary syndrome and smoking history. Other epidemiologic risk factors including tamoxifen exposure, history of breast cancer, current hormone therapy use, anticoagulant use, oral contraception use, family history of endometrial, breast or colon cancer.
Procedure: transvaginal ultrasound examination — All patients will undergo a standard transvaginal ultrasound examination followed by power Doppler endometrial vascularity assessment. After ultrasound examination, all patients will undergo endometrial sampling either through hysteroscopy or dilatation and curettage operation (D, C) or will have histopathological evaluation of biopsy specimens obtained by hysterectomy. Histopathological evaluation will serve as a gold standard for the ﬁnal diagnosis.
  Other Names: power Doppler endometrial vascularity assessment; endometrial sampling

SUMMARY:
Abnormal uterine bleeding (AUB) represents common diagnostic challenge in everyday gynecological practice. However, abnormal bleeding is a common symptom of many benign diseases and only indicates the presence of EC in 9% of postmenopausal women and 1% to 2% of premenopausal women, suggesting that many women at low risk undergo unnecessary invasive procedures to rule out cancer. The aim of the study is to create a risk-scoring model of endometrial hyperplasia and endometrial cancer.

DETAILED DESCRIPTION:
Approximately 90% of endometrial cancer (EC) cases are preceded by AUB in premenopausal or perimenopausal women or post-menopausal bleeding (PMB).Transvaginal ultrasonography(TVS) has become the first step diagnostic tool of AUB. The main advantage of ultrasound imaging is that it has high accuracy for the preoperative classiﬁcation of intra and extra uterine lesions, both benign and malignant. If increased endometrial thickness (ET) is found in women with PMB, the risk of EC increases. However, in women with type II EC, ET below 3-4 mm might also be found. Because of these limitations, ET should not be the only factor for cancer risk estimation in women with AUB.

Three-dimensional sonography and blood ﬂow vascular indices improve the diagnostic precision of the sonographic estimation of endometrial lesions. Several scoring systems using different ultrasound image characteristics were proposed to estimate the risk of EC in women with AUB including the recently proposed system" Risk of Endometrial Cancer scoring model "(REC).

Existing guidelines recommend considering clinical risk factors such as BMI, age, obesity, type II diabetes, polycystic ovary syndrome(PCOS) and use of unopposed estrogen when evaluating AUB. However, only few clinical risk prediction models have been developed.

Despite the important role of ultrasound imaging in assessment of endometrial lesions, one wonders if clinical variables can improve the diagnostic performance of risk prediction models.

The aim of the study is to create a risk-scoring model of endometrial hyperplasia and endometrial cancer using patient clinical characteristics and ultrasound image characteristics among women with abnormal uterine bleeding, and to validate the diagnostic performance of our model and to compare it's predictive value with the recently proposed REC score for EC risk stratiﬁcation.

ELIGIBILITY:
Inclusion Criteria:

women ≥40 years with pre- or perimenopausal AUB or PMB presenting to Women's Health Hospital, Department of Obstetrics and Gynecology, Faculty of medicine, Assiut University, Assiut, Egypt.

Exclusion Criteria:

* Women with a vaginal bleeding arising from a cervical, vaginal or vulvar disease.
* Patients with cervical cancer or uterine metastases.
* History of prior hysterectomy, prior pelvic radiation, endometrial sampling within the past 3 months.
* Presence of existing pregnancy.
* Women with inadequate endometrial sampling or with no histopathological diagnosis.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Eligible women presenting to Women's Health hospital with pre or peri-menopausal abnormal uterine bleeding(AUB )or Postmenopausal (PMB)will be prospectively enrolled after obtaining their informed consent. Abnormal uterine bleeding will be deﬁned by symptoms of heavy menstrual bleeding, inter-menstrual bleeding, meno-metrorrhagia, irregular menses, or other AUB among women aged ≥40 years who are not in menopause. Peri-menopausal bleeding will be defined as vaginal bleeding after 6 months of menopause after the age of 40 years. Postmenopausal status will be defined as the absence of menstruation for at least 12 months after the age of 40 years, where any pathological condition of amenorrhea is excluded.
Sampling Method: Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
prevalence of endometrial cancer, endometrial hyperplasia | 3 years
  Magnitude and prevalence of endometrial cancer, endometrial hyperplasia using a practical clinical-ultrasound based scoring system.

SECONDARY OUTCOMES:
prevalence of endometrial benign lesions | 3 years
  calculate absolute risks (prevalent risk) of endometrial benign lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke MA, Long BJ, Del Mar Morillo A, Arbyn M, Bakkum-Gamez JN, Wentzensen N. Association of Endometrial Cancer Risk With Postmenopausal Bleeding in Women: A Systematic Review and Meta-analysis. JAMA Intern Med. 2018 Sep 1;178(9):1210-1222. doi: 10.1001/jamainternmed.2018.2820. PMID 30083701
- [Background] Matteson KA, Robison K, Jacoby VL. Opportunities for Early Detection of Endometrial Cancer in Women With Postmenopausal Bleeding. JAMA Intern Med. 2018 Sep 1;178(9):1222-1223. doi: 10.1001/jamainternmed.2018.2819. No abstract available. PMID 30083765
- [Background] Pennant ME, Mehta R, Moody P, Hackett G, Prentice A, Sharp SJ, Lakshman R. Premenopausal abnormal uterine bleeding and risk of endometrial cancer. BJOG. 2017 Feb;124(3):404-411. doi: 10.1111/1471-0528.14385. Epub 2016 Oct 20. PMID 27766759
- [Background] Du J, Li Y, Lv S, Wang Q, Sun C, Dong X, He M, Ulain Q, Yuan Y, Tuo X, Batchu N, Song Q, Li Q. Endometrial sampling devices for early diagnosis of endometrial lesions. J Cancer Res Clin Oncol. 2016 Dec;142(12):2515-2522. doi: 10.1007/s00432-016-2215-3. Epub 2016 Aug 11. PMID 27515060
- [Background] Szubert S, Szpurek D, Wojtowicz A, Zywica P, Stukan M, Sajdak S, Jablonski S, Wicherek L, Moszynski R. Performance of Selected Models for Predicting Malignancy in Ovarian Tumors in Relation to the Degree of Diagnostic Uncertainty by Subjective Assessment With Ultrasound. J Ultrasound Med. 2020 May;39(5):939-947. doi: 10.1002/jum.15178. Epub 2019 Nov 29. PMID 31782548
- [Background] Gull B, Karlsson B, Milsom I, Granberg S. Can ultrasound replace dilation and curettage? A longitudinal evaluation of postmenopausal bleeding and transvaginal sonographic measurement of the endometrium as predictors of endometrial cancer. Am J Obstet Gynecol. 2003 Feb;188(2):401-8. doi: 10.1067/mob.2003.154. PMID 12592247
- [Background] Dueholm M, Hjorth IM. Structured imaging technique in the gynecologic office for the diagnosis of abnormal uterine bleeding. Best Pract Res Clin Obstet Gynaecol. 2017 Apr;40:23-43. doi: 10.1016/j.bpobgyn.2016.09.010. Epub 2016 Oct 1. PMID 27818130
- [Background] Dueholm M, Hjorth IMD, Dahl K, Pedersen LK, Ortoft G. Identification of endometrial cancers and atypical hyperplasia: Development and validation of a simplified system for ultrasound scoring of endometrial pattern. Maturitas. 2019 May;123:15-24. doi: 10.1016/j.maturitas.2019.01.017. Epub 2019 Feb 1. PMID 31027672
- [Background] Burbos N, Musonda P, Duncan TJ, Crocker SG, Morris EP, Nieto JJ. Estimating the risk of endometrial cancer in symptomatic postmenopausal women: a novel clinical prediction model based on patients' characteristics. Int J Gynecol Cancer. 2011 Apr;21(3):500-6. doi: 10.1097/IGC.0b013e31820c4cd6. PMID 21436697